CLINICAL TRIAL: NCT07403877
Title: A Phase II Randomized Controlled Trial of Neoadjuvant Immunotherapy With or Without Radiotherapy in Locally Advanced Microsatellite Instability-High/Mismatch Repair-Deficient Colorectal Cancer
Brief Title: Neoadjuvant Immunotherapy ± Radiotherapy in MSI-H/dMMR Locally Advanced Colorectal Cancer
Acronym: TORCH-OPTIMA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Chief Physician, Department of Radiation Oncology, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2025-592-4741
Record Dates: First submitted 2026-02-01; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (MSI-H)
Keywords: colorectal cancer; microsatellite instability high; mismatch repair-deficient; neoadjuvant therapy; radiotherapy; immunotherapy; locally advanced
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — Nivolumab; Ipilimumab; DEAE-Dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anti-PD-1 plus anti-CTLA-4 (Experimental): Arm A: Nivolumab 240 mg every 2 weeks (6 doses) plus ipilimumab 1 mg/kg every 3 weeks (4 doses).
  Interventions: Drug: Nivolumab; Drug: Ipilimumab (1mg/kg); Procedure: Radical surgery; Other: Watch & wait
- anti-PD-1 plus radiotherapy (Experimental): Arm B: Radiotherapy (5 Gy per fraction, total 4 fractions, delivered every 3 weeks) to the primary lesion plus nivolumab 240 mg every 2 weeks (6 doses).
  Interventions: Drug: Nivolumab; Radiation: PULSAR; Procedure: Radical surgery; Other: Watch & wait
- anti-PD-1 monotherapy (Active Comparator): Arm C: Nivolumab 240 mg every 2 weeks (6 doses).
  Interventions: Drug: Nivolumab; Procedure: Radical surgery; Other: Watch & wait

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg every 2 weeks
Drug: Ipilimumab (1mg/kg) — Ipilimumab 1 mg/kg every 3 weeks
  Arms: anti-PD-1 plus anti-CTLA-4
Radiation: PULSAR — Irradiation targeted to the primary lesion (5 Gy per fraction, total 4 fractions, delivered every 3 weeks).
  Arms: anti-PD-1 plus radiotherapy
Procedure: Radical surgery — Surgical resection will be performed in resectable cases.
Other: Watch & wait — For patients with low rectal cancer who are unable to preserve the anal sphincter, a watch-and-wait (WW) strategy can be considered if a clinical complete response (CR) is achieved.

SUMMARY:
This phase II clinical trial evaluates the efficacy and safety of three neoadjuvant regimens in patients with locally advanced microsatellite instability-high/mismatch repair-deficient (MSI-H/dMMR) colorectal cancer (CRC): 1) Regimen A: Dual immune checkpoint blockade with nivolumab plus ipilimumab. 2) Regimen B: Nivolumab plus radiotherapy. 3) Regimen C: Nivolumab monotherapy. The primary objectives are to determine whether: 1) Dual immune checkpoint blockade (Regimen A) is superior to nivolumab monotherapy (Regimen C); and 2) Immunotherapy plus radiotherapy (Regimen B) is superior to nivolumab monotherapy (Regimen C). Methods: Participants will be randomized in a 1:1:1 ratio to one of the three arms. For patients with resectable tumors, surgical resection will be performed. In patients with low rectal cancer and poor prospects for sphincter preservation, a watch-and-wait (WW) strategy is an option if a clinical complete response (CR) is achieved following neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed primary colorectal adenocarcinoma.
2. Radiographic assessment showed a stage II-III based on AJCC Stage 8th ed.
3. At least 18 years old.
4. MSI-H or dMMR.
5. The Eastern Cooperative Oncology Group performance status (ECOG PS) score is 0 or 1.
6. Physical state or organ function can tolerate the planned treatment of the study protocol.
7. Agreed to sign written informed consent before recruitment.

Exclusion Criteria:

1. Previously received any antitumor therapy for the disease under study, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.
2. Pregnancy or breastfeeding women.
3. History of other malignancies within 5 years.
4. Serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
5. Immunodeficiency disease or long-term using of immunosuppressive agents.
6. Allergic to any component of the therapy.
7. Any other condition or disease that is not suitable to take the therapy included in the protocol.
8. Concurrent participation in another clinical study, unless participating in an observational (non-interventional) clinical study or in the survival follow-up phase of an interventional study.
9. Received any investigational drug or device treatment within 4 weeks prior to initial administration of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete regression (CR) rate | 1 month after surgery or the completion of neoadjuvant therapy
  Proportion of patients achieving either clinical CR (and undergoing WW) or pathological CR (confirmed by pathology) among all evaluable patients.

SECONDARY OUTCOMES:
R0 resection rate | 1 month after surgery
  Proportion of patients who achieve R0 resection.
Objective response rate (ORR) | 6 months after the enrollment of the last subject
  Proportion of patients with complete response (CR) or partial response (PR) to preoperative multimodal therapy. ORR will be evaluated using RESIST1.1 by CT/MRI of the chest, abdomen, and pelvis.
Event-free survival (EFS) | 36 months after the enrollment of the last subject
  The EFS was defined as the time from randomization to the first determination of inoperable disease progression, postoperative local recurrence or distant metastasis, tumor regrowth, or death from any cause, whichever occurs first.
Overall survival (OS) | 36 months after the enrollment of the last subject
  OS is defined as the time interval from enrollment to death of any reason or censoring.
Toxicities | From the time of enrollment, assessed up to 28 days after the last dose of study therapy
  Number of participants with treatment-related adverse events (TrAEs) reported between the first dose and 28 days after the last dose of study therapy as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Surgical morbidity | During or one month after surgery
  Surgery related adverse events (SRAEs) refer to complications which happen during or one month after surgery. Severe complications after surgery will be documented and classified by Clavien-Dindo classification, such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, and incision complications (infection, bleeding, rupture).
Surgical mortality | During or one month after surgery
  Death from any cause within 30 days of the date of surgery will be considered a surgical mortality death.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No